CLINICAL TRIAL: NCT04892745
Title: Impact of Hemodialysis on Cutaneo-muscular Electrical Impedance
Acronym: H-ICMUS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210098; 2020-A03337-32 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-04-16; First posted 2021-05-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hemodialysis
Keywords: hemodialysis; electrical impedance; subcutaneous impedancemetry; cutaneo-muscular impedancemetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of this pilot study aims to describe the modifications of subcutaneous impedancemetry induced by dialysis.

As secondary objectives, the study aims to 1) describe the modifications of cutaneo-muscular impedancemetry induced by dialysis. 2) describe the relationship between modifications of subcutaneous impedancemetry induced by dialysis and - technical conditions of dialysis; - volemic parameters of dialysis; - evolution of liquid compartments in organism during dialysis; - volemic events or neuromuscular events. 3) describe the relationship between modifications of cutaneo-muscular impedancemetry induced by dialysis and 1) describe the modifications of cutaneo-muscular impedance induced by dialysis. 2) describe the relationship between modifications of subcutaneous impedancemetry induced by dialysis and - technical conditions of dialysis; - volemic parameters of dialysis; - evolution of liquid compartments in organism during dialysis; - volemic events or neuromuscular events.

DETAILED DESCRIPTION:
The study will be realized in dialysis facility of Ambroise Paré hospital, APHP. The duration of enrollment of subjects will be 3 months, each enrolled patient will has 2 or 3 week's follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient ⩾ 18 years;
* Patient undergoing chronic dialysis in hemodialysis facility of Ambroise Paré hospital;
* Patient has been informed and given no-opposition for participating to the study.

Exclusion Criteria:

* Patient with a pacemaker or an implantable cardioverter defibrillator;
* Patient under guardianship or curatorship;
* Foreign patient under french AME scheme.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering chronic renal failure and undergoing chronic hemodialysis in Ambroise Paré hospital.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Electrical parameters of subcutaneous impedancemetry | at the end of study, up to 4 months
  Electrical parameter extracellular resistance (Re) will be assessed.

SECONDARY OUTCOMES:
Cutaneo-muscular impedancemetry assessement | at the end of study, up to 4 months
  Cutaneo-muscular impedancemetry will be assessed by extracellular resistance (Re).
Whole body impedancemetry assessement | at the end of study, up to 4 months
  Whole body impedancemetry will be assessed by Re.
Incidence of volemic or neuromuscular events | at the end of study, up to 4 months
  Incidence of volemic or neuromuscular events during the session, such as:
  * peridialytic hypotension,
  * crampses.

CONTACTS AND LOCATIONS:
Overall Officials: Marie ESSIG, MD, PhD, Principal Investigator — Service de Néphrologie, Hôpital Ambroise Paré, APHP
Locations (1):
- Service de Néphrologie, Hôpital Ambroise Paré, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No